CLINICAL TRIAL: NCT01836783
Title: A Prospective Study of Bone Augmentation Techniques in Extraction Sockets
Brief Title: Bone Augmentation Techniques in Extraction Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: BioDlogics (Industry)
Responsible Party: Principal Investigator, Maninder Kaur, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amnio-12
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Tooth Loss
Keywords: Allograft; Amnion Allograft
MeSH Terms: conditions — Tooth Loss | interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amnion Allograft (Experimental): Atraumatic tooth extractions and amnion allograft procedures
  Interventions: Other: Amnion Allograft
- Allograft (Active Comparator): Atraumatic tooth extractions and allograft procedures
  Interventions: Other: Allograft

INTERVENTIONS:
Other: Amnion Allograft — Atraumatic extraction and grafting procedures will be followed by insertion of a dental implant into the grafted area at week-8. The implant will be restored and be monitored for 24 months post-insertion. Two special dental cone-beam CT images (pre-baseline and week-7) and a minimum of 6 intraoral radiographs will be taken during the study
  Arms: Amnion Allograft
Other: Allograft — Atraumatic extraction and grafting procedures will be followed by insertion of a dental implant into to the grafted area at week-8. The implant will be restored and be monitored for 24 months post-insertion. Two special dental cone-beam CT images (pre-baseline and week-7) and a minimum of 6 intraoral radiographs will be taken during the study
  Arms: Allograft

SUMMARY:
The study will compare the density and strength of regenerated bone in extraction sockets after being grafted with two different materials: Bone Allograft and Bone Allograft with Amnion.

The investigators hypothesize that sockets grafted with the Amnion graft will exhibit enhanced healing patterns and will accelerate the formation of regenerated bone in the grafted areas.

DETAILED DESCRIPTION:
The amniotic allograft is a cryopreserved allograft tissue matrix derived from human placental tissues recovered from live healthy donors. Amniotic tissue is an abundant source of collagen which provides an extracellular matrix to act as a natural scaffold for cellular attachment in the body; collagen provides a structural tissue matrix that facilitates cellular migration and proliferation in-vivo. The product is developed using proprietory techniques by BioDlogics, LLC. The amniotic allograft growth factors are thought to enhance formation of a supportive scaffold for regeneration, to facilitate interactions between cell types, and to influence anti-inflammatory, anti-microbial and immuno-privilege activities.

Atraumatic extractions and socket grafts will be performed. Dental implants will be inserted into the grafted areas 8 weeks post-graft. The implants will be restored and followed for 24 months post-insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Be a registered University of Alabama at Birmingham (UAB) dental school patient
2. Existence of one or more non-adjacent teeth in the aesthetic zone that are scheduled for extraction
3. Healthy enough to undergo the proposed therapy
4. Demonstrated willingness to comply with study directions and time-line
5. Able to consent for themselves
6. Able to read and understand the informed consent form -

Exclusion Criteria:

1. Pregnant or lactating at the time of enrollment
2. Previous Malignant neoplasm
3. Known hypersensitivity to bone grafting materials
4. Know hypersensitivity to titanium
5. Any medical of medication that in the opinion of the investigators may adversely affect bone healing
6. Any indication of an inability to make autonomous decisions -

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maninder Kaur, BDS MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amnion Allograft | Allograft
Started | 10 | 12
Completed | 10 | 10
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amnion Allograft | Allograft | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Hard Tissue Composition
Description: A biopsy will be harvested from each grafted-site and sent to a laboratory for histological and histomorphometric analysis
Time Frame: baseline to week-8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Amnion Allograft | Allograft
Number analyzed (Participants) | 10 | 10
mm | 35.82 (13.16) | 31.76 (20.03)

2. Secondary Outcome: Changes in Soft Tissue Healing
Description: Clinical examination utilizing photographic data and imaging analysis software
Time Frame: baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: square millimeters
Arm/Group | Amnion Allograft | Allograft
Number analyzed (Participants) | 10 | 10
square millimeters | 12.41 (8.74) | 12.79 (7.7)

3. Secondary Outcome: Changes in Soft Tissue Healing
Description: Clinical examination utilizing photographic data and imaging analysis software
Time Frame: 2 weeks to 7 weeks
Measure: Mean (Standard Deviation); unit: square millimeters
Arm/Group | Amnion Allograft | Allograft
Number analyzed (Participants) | 10 | 10
square millimeters | 0.87 (1.44) | 1.78 (3.06)

ADVERSE EVENTS:
Time Frame: baseline to week 7
Arm/Group | Amnion Allograft | Allograft
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT01836783/Prot_SAP_000.pdf